CLINICAL TRIAL: NCT05608499
Title: Efficacy and Safety of Duobrii in the Management of Acne Keloidalis Nuchae (AKN)
Brief Title: Duobrii Treatment of Acne Keloidalis Nuchae (AKN)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis did not show any significant differences between groups
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Principal Investigator, Benjamin Ungar, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO-22-0955
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Acne Keloidalis Nuchae; AKN
MeSH Terms: conditions — Acne Keloid | interventions — halobetasol; tazarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Duobrii (Experimental): Duobrii is the study treatment drug. Bryhali will only be used as a rescue treatment - in case of irritation with Duobrii.
  Interventions: Drug: Duobrii; Drug: Bryhali
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duobrii — topical contains active drug lotion, once daily for 4 weeks then twice daily for 8 weeks
  Other Names: halobetasol propionate and tazarotene
  Arms: Duobrii
Drug: Placebo — Topical does not contain active properties of study drug
  Arms: Placebo
Drug: Bryhali — Bryhali will only be used as a rescue treatment - in case of irritation with Duobrii. Bryhali lotion once daily up to 12 weeks only if Duobrii is not tolerated.
  Other Names: halobetasol propionate
  Arms: Duobrii

SUMMARY:
Acne keloidalis nuchae (AKN) is one of the chronic forms of scarring folliculitis, affecting predominantly the occipital scalp, seen mostly in men of African descent. Duobrii has the advantage of being the only high potency topical steroid-retinoid combination approved by the FDA with dermatologic indication. Researchers are proposing the off-labeled use of Duobrii for the management of early-mild AKN. The research team hypothesizes that subjects will experience significant clinical improvement in lesion counts. Patients will be followed with visits scheduled at baseline, 4 weeks, 8 weeks, and 12 weeks. During these in-clinic visits, there will be surveys regarding the severity of AKN symptoms, photographs, and clinical assessments.

DETAILED DESCRIPTION:
Acne keloidalis nuchae (AKN) is one of the chronic forms of scarring folliculitis, affecting predominantly the occipital scalp, seen mostly in men of African descent. Duobrii has the advantage of being the only high potency topical steroid-retinoid combination approved by the FDA with dermatologic indication. Researchers are proposing the off-labeled use of Duobrii for the management of early-mild AKN. The research team hypothesizes that subjects will experience significant clinical improvement in lesion counts.

Enrolled participants will be instructed to apply placebo (n=10) vs. active (n=20) to affected area of the occipital scalp for 4 weeks once a day (label use). Each application will be approximately 1g. Following the 4 weeks, participants will be instructed to increase application to twice daily (BID; off-label; at least 8 hours apart) for one week. Investigators will conduct a phone visit on week 5 to discuss any potential side effects with this increased dose. If tolerated, this BID regimen will be carried throughout the length of the study. If BID is not tolerated (if irritation occurs), then Bryhali will be used as a "rescue treatment" once daily for 1 week before the subject returns to BID treatment with Duobrii. If irritation recurs, subjects will be instructed to alternate Duobrii and Bryhali (ie Duobrii BID one day, followed by Bryhali QD the next day, Duobrii BID the next, and so on). Alternating topical steroid use and stepping down topical steroid strength have been known to reduce lesion count in AKN.3 If irritation continues to persist, then participants will be instructed to use Bryhali QD for five days a week and Duobrii BID two days a week. If participants still experience irritation with this regimen, then subjects will be transitioned entirely to Bryhali QD for the remainder of the study. In case of clearance earlier than the end of the study, participants will be instructed to continue their respective regimen to completion of the study. Gentle hair care regimen will be recommended for duration of the length of the study; with unscented shampoo & conditioner (such as Head & shoulder) and Vaseline to scalp as moisturizer to minimize risk of contact dermatitis. In addition, patients will be instructed to postpone any form of hair coloring or chemical hair processing until after the study is over.

Participants will be followed with visits scheduled at baseline, 4 weeks, 8 weeks and 12 weeks. At each visit, participants will complete surveys regarding the severity of AKN's associated symptoms (pain, pruritus, burning etc.) as well as the dermatology quality of life index (DLQI) and numerical rating scale (NRS) surveys (Appendix B&D). In addition, photographs will also be obtained for global assessment and lesion count will be performed. The investigator will assess the treatment area for any dyspigmentation and document the % area affected within the treatment area at each visit. Tape strips will also be collected from lesional (occipital scalp) and non-lesional (frontal scalp) at Baseline and Week 12. There will be a phone call visit at week 5 to assess tolerance of medication increase and a safety follow-up visit at Week 14. Statistical analysis will be performed. Throughout the length of the study, any adverse events (AEs) related to the treatment will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least 18 years of age
* Subject is able to provide written informed consent and comply with the requirements of this study protocol
* Subjects have AKN class I or II (less than 6.5 cm in width)
* Subjects who are women of childbearing potential (WOCBP) must have a negative urine pregnancy test at screening and must be practicing an adequate and medically acceptable method of birth control for at least 30 days prior to Day 0 and at least 6 months after the last dose of study. Acceptable methods of birth control include:

  * intrauterine device (IUD) oral;
  * transdermal;
  * implanted or injected hormonal contraceptives (must have been initiated at least 1 month before entering the study);
  * tubal ligation;
  * abstinence;
  * barrier methods with spermicide.
* If not of child-bearing potential, subjects must have:

  * a sterile or vasectomized partner;
  * have had a hysterectomy;
  * a bilateral oophorectomy or be clinically diagnosed infertile;
  * or be in a menopausal state for at least a year.
  * Subject is judged to be in good general health as determined by the principal investigator.

Exclusion Criteria:

* unable to understand and provide written consent
* Have received prior intralesional steroids for AKN within the past 6 months
* Are using topical steroids or topical medications on their scalp within 4 weeks
* Have used Duobrii on the scalp for AKN or other scalp disorders
* Subject is pregnant or breastfeeding
* Use of prior systemic medication for AKN or acne (doxycycline or isotretinoin) or hair loss in the last 6 months
* Currently using topical minoxidil or prior use within the past 3 months
* Have a history of other or other active scalp/hair disease or other forms of or other forms of alopecia
* Are on systemic steroids or other immunosuppressants
* Have a history of auto-immune disease, thyroid disorder, or hypersensitivity to steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin N Ungar, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. Aggregated data will be discussed in the final published article.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duobrii | Placebo
Started | 10 | 5
Completed | 9 | 4
Not Completed | 1 | 1
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duobrii | Placebo | Total
Number analyzed (Participants) | 10 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (10.23) | 32 (6.67) | 33 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Lesion Count
Description: Change in Lesion Count between baseline and Week 12
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | Duobrii | Placebo
Number analyzed (Participants) | 10 | 5
lesion count | 3.89 (15.28) | -5.5 (15.78)

2. Secondary Outcome: Changes in Pain Rating Scale
Description: Changes in Pain Rating Scale as compared to baseline. Full scale is 0-10, where higher scores indicate greater severity of AKN pain symptoms.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Duobrii | Placebo
Number analyzed (Participants) | 10 | 5
score on a scale | 1 (2.45) | -0.25 (0.957)

3. Secondary Outcome: Changes in Itch Rating Scale
Description: Changes in Itch Rating Scale as compared to baseline. Full scale is 0-10, where higher scores indicate greater severity of AKN itch symptoms.
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Duobrii | Placebo
Number analyzed (Participants) | 10 | 5
score on a scale | 0.333 (2.12) | -3 (1.83)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Duobrii | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5
Other Adverse Events (participants affected / at risk) | 4/10 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Duobrii (N=10) | Placebo (N=5)
Scalp Irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Scalp Irritation /Erythema at site of AKN (Skin and subcutaneous tissue disorders) | 1 | 0
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT05608499/Prot_SAP_001.pdf
  • Informed Consent Form (2024-07-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT05608499/ICF_000.pdf